CLINICAL TRIAL: NCT07107516
Title: Safety and Immunogenicity of PanChol, a Novel Live Attenuated Oral Cholera Vaccine, in Zambia Adults
Brief Title: Phase 1b Ascending Dose Study of PanChol in Healthy Volunteers
Acronym: PanChol
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Centre for Infectious Disease Research in Zambia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PanChol 101
Record Dates: First submitted 2025-07-30; First posted 2025-08-06 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Cholera Vaccination Reaction
Keywords: cholera; vaccine; safety
MeSH Terms: conditions — Cholera

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- cohort 2a (Experimental): The PanChol vaccine will be given at a dose of 2 x 10^7 CFU in this arm
  Interventions: Biological: PanChol
- cohort 2b (Experimental): The PanChol vaccine will be given at a dose of 2 x 10^8 CFU in this arm
  Interventions: Biological: PanChol
- cohort 2c (No Intervention)

INTERVENTIONS:
Biological: PanChol — Panchol is a novel live attenuated oral cholera vaccine. It is the first vaccine created with the variant El Tor background that is predominant in the world today. The vaccine has ten different genetic modifications to minimize reactogenicity but maintain the ability to colonize the intestine.
  Arms: cohort 2a; cohort 2b

SUMMARY:
Cholera is a serious diarrheal disease that can be fatal within hours of onset. The current available cholera vaccines to prevent the disease are not very effective. Panchol is a new oral cholera vaccine that may be an improvement over the currently available vaccines in use. The goal of this study is to learn safety of this new oral cholera vaccine and the body's immune response to the vaccine.

The researchers will compare the PanChol vaccine to placebo to see the side effects experienced in participants.

The participants will be adults aged between 18 and 55 years and they will be required to:

1. Be admitted to hospital until they stop passing the cholera vaccine in their stool. During admission, all side effects will be recorded by the researchers.
2. After discharge, the participants will visit the research site every month for 3 months with an optional visit at the 4th month for the researchers to assess the participants' general health.

ELIGIBILITY:
Inclusion Criteria:

1. Must have given written informed consent (signed and dated) and any other authorizations required by local law and be able to comply with all study requirements.
2. Healthy adults aged from 18 to 55 years old.
3. Considered healthy, as judged by the clinical investigator, according to medical history, physical examination, vital signs, screening laboratories, and medication history.
4. Capable of understanding, consenting, and complying with the entire study protocol including the inpatient period.
5. Female participants must be non-pregnant and non-lactating and either

   1. surgically sterile (history of bilateral ligation, bilateral salpingectomy, bilateral oophorectomy, total hysterectomy) or postmenopausal (defined as amenorrhea for at least 12 consecutive months before screening without an alternative medical cause)
   2. be of child-bearing potential and practicing an acceptable method of contraception or abstaining from all activities that could result in pregnancy for at least 28 days before vaccination until 3 months after receiving the investigational product.

Acceptable methods of contraception include barrier methods (such as condom, diaphragm, or cervical cap used in conjunction with spermicide), intrauterine device, hormonal contraception (that may be taken or administered by oral, intravaginal, transdermal, subdermal or IM route), vasectomized partner (the vasectomized partner should be the sole partner for that participant)

Exclusion Criteria:

1. Confirmed or suspected immunosuppressive condition, as a result of a disease (e.g., primary immune deficiency, malignancy, HIV infection) or have taken any systemic immunosuppressive therapy within 6 months of enrollment.
2. Pregnant or lactating women.
3. History of gastrointestinal (GI) disorder, such as previous major GI surgery, malabsorption, or any chronic GI disorders that would interfere, according to the investigator, with the IP.
4. Acute GI or febrile illness within 7 days of enrollment.
5. Have any acute or chronic medical condition that, in the opinion of the investigator, would make vaccination unsafe or interfere with the evaluation of immune response to study vaccination.
6. History of cholera vaccination.
7. History of cholera infection.
8. Abnormal stool pattern, defined as < 3 or >21 stools per week.
9. Allergy or intolerance to PanChol or placebo component (sodium bicarbonate, lactose, ascorbic acid)
10. Use of any systemic antibiotics within 1 month of PanChol administration.
11. Receipt of a live vaccine in the previous 4 weeks or planned in the 4 weeks following enrollment.
12. Receipt of a killed or subunit (non-live) vaccine in the previous 2 weeks or planned in the 2 weeks following enrollment.
13. Individuals who do not speak English
14. Childcare workers with direct contact with children ≤ 2 years of age
15. Individuals whose occupation involves handling of food
16. Healthcare workers who have direct contact with patients who are immunodeficient, HIV-positive, or have an unstable medical condition
17. Use laxatives regularly
18. Have diarrhea within 48 hours before enrollment
19. Have a history of hypersensitivity to any of the tetracyclines
20. Have a history of hypersensitivity to streptomycin or any aminoglycoside due to the known cross-sensitivity of patients to drugs in this class.
21. Individuals who have a household member who are immunodeficient, HIV-positive, or have an unstable medical condition.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
vaccine safety | 14 days after vaccination
  The incidence of solicited and unsolicited adverse events, including serious adverse events, following PanChol vaccination

SECONDARY OUTCOMES:
immunogenicity | 180 days after vaccination
  The seroconversion (4-fold rise titer over baseline) of the vibriocidal titers to both Inaba and Ogawa V. cholerae between pre- and post-vaccination with PanChol.
vaccine stool shedding | 8 days after vaccination
  Stool shedding of PanChol organisms using quantitative and qualitative stool cultures

OTHER OUTCOMES:
exploratory- serum antibody changes | 180 days after vaccination
  Changes of IgG, IgA, and IgM antibodies targeting Inaba- and Ogawa-specific polysaccharides, CT-B and TCP.
exploratory- IgA and IgG secreting cell responses | 180 days after vaccination
  Changes of IgA- and IgG-antibody secreting cell responses (ALS/plasmablast responses) and the memory B cell (MBC) response.
Exploratory- Microbiome modification | 180 days after vaccination
  Stool microbiota modification according to 16S rRNA sequencing and/or metagenomic sequencing

CONTACTS AND LOCATIONS:
Locations (1):
- CIDRZ Matero clinical reseach site, Lusaka, Lusaka Province, Zambia

IPD SHARING:
Plan to Share IPD: Undecided